CLINICAL TRIAL: NCT06873152
Title: Improvement of Operating Room Efficiency in the Extraction of Bilateral Third Molar Surgery Under Narcosis Using Enhanced Preoperative Preparation and a Dedicated Operating Room Team: a Randomised Controlled Trial (PREPARE-study)
Brief Title: Improvement of Operating Room Efficiency in Bilateral Wisdom Teeth Surgery
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Prof Dr, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/007
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Third Molars Extraction
Keywords: operation room efficiency; third molar surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): The operation room team will consist of a randomly planned team which may also comprise nurse trainees and/or anesthesiology residents.
  At arrival in the operating theatre, all patients will be placed in the supine position and receive full standard monitoring (non-invasive blood pressure monitoring, electrocardiographic monitoring, and peripheral O2 saturation monitoring). Furthermore, they will receive an intravenous access with 0.9% sodium chloride infusion and will be administered clindamycine 900mg IV.
  Interventions: Procedure: Control preoperative program
- Experimental group (Experimental): All patients planned on an experimental stomatology program day will receive an intravenous access with 0.9% sodium chloride infusion at the ambulatory ward and will be administered clindamycine 900mg IV 30 minutes before the start of surgery.
  During an experimental stomatology program day, the OR team will consist of 2 very well-trained OR nurses who are exclusively dedicated to the maxillofacial surgery department and a highly experienced anesthesiologist who also has frequent exposure to surgical maxillofacial interventions programs. Nurse trainees and/or anesthesiology residents will not be planned in the stomatology OR on experimental days.
  Interventions: Procedure: Advanced preoperative program

INTERVENTIONS:
Procedure: Control preoperative program — Patients will undergo a control preoperative program with no enhances preparation when undergoing bilateral third molar extraction
  Arms: Control group
Procedure: Advanced preoperative program — Patients will undergo an comprehensive program including enhanced preoperative preparation and a dedicated operating room team when undergoing bilateral third molar extraction
  Arms: Experimental group

SUMMARY:
This study aims to assess and compare the implementation of this comprehensive program in patients undergoing bilateral third molar extraction on OR and hospital efficiency and patient experience. The investigators hypothesize that this comprehensive program will be superior in terms of OR efficiency compared to "business as usual".

DETAILED DESCRIPTION:
Operating room (OR) efficiency is an important parameter for hospital cost-efficiency since the OR is a high-cost unit. Time is the most valuable resource of an OR. For example, in fiscal year 2014 for California's acute care hospitals, cost attributable to fixed overhead to utilize an OR was an estimated $20 per minute. When factoring in physician and nursing staff, the mean cost of operating room time in the ambulatory setting was $36 per minute.

In that regard, the nonoperative time (NOT) defined as the time between surgical completion of the previous patient and skin incision on the following patient is an important parameter. The NOT can be calculated as the sum of Anesthesia induction time (IT), the emergence time (ET), and the turnover time (TOT) and has the potential to improve or reduce operating room efficiency substantially, especially in short-duration surgery programs. On the other hand, mismanagement of NOT may have negative impact on OR efficiency and surgeon's, patient's, and staff's satisfaction.

In that regard, IT of general anesthesia can be strongly prolonged due to difficulties in obtaining venous access. ET from general anesthesia that starts after completion of the surgical procedure and the cessation of anesthetic delivery until extubation is largely under the control of the anesthetist. It can be influenced by anesthetic agent choice, dose, and dose duration and moreover the risk of prolonged ET is inversely related with the anesthesia resident training duration. TOT is defined as the time from when the patient's bed exited the OR to the time when the next patient's bed entered the OR and is mostly influenced by the efficiency of the housekeeping staff to clean the OR and the nursing team to prepare the OR for the next patient.

Bilateral third molar surgery is one of the most commonly performed short-duration procedures performed in an ambulatory setting. Dental surgery performed under general anesthesia is associated with minimized anxiety and high patient satisfaction levels. Therefore, general anesthesia is recommended in patients with severe anxiety or pronounced vomiting reflex and in patients undergoing bilateral third molar surgery.

To improve OR efficiency during bilateral third molar surgery under general anesthesia, the investigators have developed a comprehensive program including enhanced preoperative preparation of patients, the development of a procedure-specific anesthesia protocol and the formation of a dedicated operating room team. Enhanced preoperative preparation includes preoperatively performing intravenous cannulation and administration of intravenous antibiotics on the ambulatory ward. In the anesthesia protocol, only short or very short acting agents are selected and the dedicated operating room team consists of 2 very well-trained OR nurses and a highly experienced anesthesiologist who all have frequent exposure to surgical stomatology programs.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-60 years
* ASA I- III
* BMI ≤ 40 kg/m2
* Patient is willing to give informed consent
* Patient is scheduled for wisdom teeth surgery

Exclusion Criteria:

* The inability to understand to the study design
* Refusal to participate in the trial

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of total operation room stay time | on day of surgery, day 0
  Evaluation of the Total Operation room (OR) stay time defined as departure time from the OR minus arrival time in the OR

SECONDARY OUTCOMES:
Evaluation of the surgical time | on day of surgery, day 0
  Evaluation of the Surgical time (ST) defined as the time from application of dressings and incision to surgical completion
Evaluation of Anesthesia induction time | on day of surgery, day 0
  Evaluation of Anesthesia induction time (IT) defined as time interval between arrival to the OR and patient handover to surgical team.
Evaluation of emergence time | on day of surgery, day 0
  Emergence time (ET) defined as the time interval between end of surgery and patient wheeled out of the OR
evaluation of turnover time | on day of surgery, day 0
  turnover time (TOT) defined as the time from when the patient's bed exited the OR to the time when the next patient's bed entered the OR
Evaluation of non operative time | on day of surgery, day 0
  - Nonoperative time (NOT) defined as the time between surgical completion of the previous case and skin incision on the following case.
Evaluation of pain | baseline, 4, 8 and 24hours after surgery
  - Mean postoperative pain intensity at rest measured by an 11-point Numeric Rating Scale (NRS) (with 0 no pain and 10 extreme pain) at baseline, 4, 8 and 24 hours after surgery
Evaluation of hospital length of stay | on day of surgery, day 0
  Evaluation of hospital length of stay in hours
Evaluation of time to be fit for discharge | on day of surgery, day 0
  - Time to be fit for hospital discharge after the end of surgery as defined by reaching all of the following criteria:
  * Oral pain medication only
  * Independent walking
  * No PONV
  * Bowel movement
  * Oral Intake
  * Hemodynamically (90% of baseline BP, HR in 90% of normal range) and respiratory stable (no need for extra oxygen)
  * No drains or urinary catheters
Evaluation of patient satisfaction | one day after the surgery, day 1
  General patient satisfaction with perioperative anesthesia and analgesia: this will be evaluated by telephone call at postoperative day (POD) 1 by the study assistant with a 10-point Likert Scale with 1 being extremely dissatisfied and 10 being extremely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium